CLINICAL TRIAL: NCT02640833
Title: A Phase 1b/2 Study of Duvelisib and Venetoclax in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia, Small Lymphocytic Lymphoma, or Indolent or Aggressive Non-Hodgkin Lymphoma, Who Have Not Previously Received a Bcl-2 or PI3K Inhibitor
Brief Title: A Study of Duvelisib and Venetoclax in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia, Small Lymphocytic Lymphoma, or Indolent or Aggressive Non-Hodgkin Lymphoma, Who Have Not Previously Received a Bcl-2 or PI3K Inhibitor
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study Stopped
Sponsor: AbbVie (Industry)
Collaborators: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-330; 2015-003302-16 (EudraCT Number)
Record Dates: First submitted 2015-12-23; First posted 2015-12-29 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Non-Hodgkin Lymphoma
Keywords: Refractory Lymphoma; Relapsed Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma; Leukemia | interventions — duvelisib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duvelisib+Venetoclax (Experimental)
  Interventions: Drug: Duvelisib; Drug: Venetoclax

INTERVENTIONS:
Drug: Duvelisib — Duvelisib will be taken continuously. This is a defining dose study, therefore the dose of Duvelisib may change.
Drug: Venetoclax — Venetoclax will be taken continuously. This is a defining dose study, therefore the dose of Venetoclax will change.

SUMMARY:
This study is designed to assess the safety, pharmacokinetics, drug-drug interactions, and determine the recommended Phase 2 doses of co administered Duvelisib and Venetoclax in participants with relapsed or refractory chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma, or indolent or aggressive non-Hodgkin lymphoma, who have not previously received a Bcl-2 or Phosphoinositide 3-kinase (PI3K) inhibitor. The Phase 2 portion of the study will preliminarily evaluate efficacy, and expand the toxicity evaluation.

ELIGIBILITY:
Inclusion Criteria: -

Subject must have either • Relapsed or refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (for Waves 2 or 3)

* Subject has evaluable disease and requires treatment in the opinion of the investigator.
* Subject must have relapsed following or be refractory to ≥ 1 standard treatments such as fludarabine based regimens (F, FC, FR, FCR), alkylator (chlorambucil, bendamustine) based regimens, or Bruton's Tyrosine Kinase inhibitor (Ibrutinib).

Or

• Relapsed or refractory indolent Non-Hodgkin Lymphoma or aggressive Non-Hodgkin Lymphoma (for Waves 1, 2, or 3, unless otherwise indicated)

* Subject must have histologically documented diagnosis of a Follicular Lymphoma or Marginal Zone Lymphoma.
* Subject must have histologically documented diagnosis of a Diffuse Large B-cell Lymphoma (excluding Richter's Transformation), Non-cutaneous T-Cell Lymphoma, or Mantle Cell Lymphoma (MCL) (MCL Wave 3 only)
* Subject has evaluable disease and requires treatment in the opinion of the investigator.
* Subject must have relapsed following or be refractory to ≥ 1 standard treatments such as R-CHOP, R-CVP, bendamustine, lenalidomide-rituximab, or fludarabine-based regimens.

  * Subject has an Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to 2.
  * Subject must have adequate bone marrow independent of growth factor support per local laboratory reference range at Screening.
  * Subject must have adequate coagulation, renal, and hepatic function, per laboratory reference range at Screening.
  * NHL subjects who have a history of an autologous stem cell transplant (e.g., bone marrow) must be > 6 months post-transplant (prior to the first dose of study drug) and must not require any growth factor support.

Exclusion Criteria:

* Subject has been previously treated with a Bcl-2 or PI3K inhibitor.
* Subject is a candidate to receive another second-line therapy approved for usage by the local Health Authority.
* Subject is appropriate for a stem cell transplant or has undergone an allogeneic stem cell transplant.
* Subject has received any of the following within 14 days or 5 drug half-lives (whichever is shortest) prior to the first dose of duvelisib or venetoclax, or has not recovered to less than Grade 2 clinically significant adverse effect(s)/toxicity(s) of the previous therapy:

  * Any anti-cancer therapy including chemotherapy or radiotherapy;
  * Investigational therapy, including targeted small molecule agents.
* Subject has received biologic agents (e.g., monoclonal antibodies) for anti-neoplastic treatment within 30 days prior to first dose of duvelisib or venetoclax.
* Subject has received live or live attenuated vaccines within 6 weeks prior to first dose of duvelisib or venetoclax.
* Subject has received the following within 7 days prior to the first dose of duvelisib or venetoclax:

  * Steroid therapy for anti-neoplastic treatment;
  * Strong and Moderate CYP3A inhibitors;
  * Strong and Moderate CYP3A inducers;
  * Chronic immunosuppressants, other than corticosteroids given at daily dose < 20 mg prednisone equivalent for ITP or AIHA.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2020-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | From participant's first dose until 30 days after participant's last dose of study drug; up to 2 years following last participant first dose
  Participants will be monitored for clinical and laboratory evidence of adverse events throughout the study.
Maximum observed plasma concentration (Cmax) of duvelisib | Blood samples will be taken at 0 (pre-dose) 1,2,4,6,8,10 and 12 hours post-dose on Cycle 1 Day 14 and Day 22 for second and third dose levels.
  The highest concentration that a drug achieves in the blood after administration in a dosing interval.
Maximum observed plasma concentration (Cmax) of venetoclax | Blood samples will be taken at 0 (pre-dose) 1,2,4,6,8,10, 12 and 24 hours post-dose on Cycle 1 Days 7 and 14, and Day 22 for second and third dose levels.
  The highest concentration that a drug achieves in the blood after administration in a dosing interval.
Time to maximum observed plasma concentration (Tmax) of duvelisib | Blood samples will be taken at 0 (pre-dose) 1,2,4,6,8,10 and 12 hours post-dose on Cycle 1 Day 14 and Day 22 for second and third dose levels.
  The time at which the maximum plasma concentration (Cmax) is observed.
Time to maximum observed plasma concentration (Tmax) of venetoclax | Blood samples will be taken at 0 (pre-dose) 1,2,4,6,8,10,12 and 24 hours post-dose on Cycle 1 Days 7 and 14, and Day 22 for second and third dose levels.
  The time at which the maximum plasma concentration (Cmax) is observed.
Area under the plasma concentration-time curve from time 0 to 12 hours post-dose (AUC12) of duvelisib | Blood samples will be taken at 0 (pre-dose) 1,2,4,6,8,10 and 12 hours post-dose on Cycle 1 Day 14 and Day 22 for second and third dose levels.
  The area under the plasma concentration-time curve over a 12-hour dose interval
Area under the plasma concentration-time curve from time 0 to 24 hours post-dose (AUC24) of venetoclax | Blood samples will be taken at 0 (pre-dose) 1,2,4,6,8,10,12 and 24 hours post-dose on Cycle 1 Days 7 and 14, and Day 22 for second and third dose levels.
  The area under the plasma concentration-time curve over a 24-hour dose interval
Recommended phase two dose (RPTD) of Duvelisib in combination with venetoclax | Minimum first cycle of dosing (28 days)
Recommended phase two dose (RPTD) of Venetoclax in combination with duvelisib | Minimum first cycle of dosing (28 days)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Measured up to 2 years after the last participant has enrolled in the study
  Progression-free survival will be defined as the number of days from the date of study drug start to the date of documented disease progression, relapse of death due to any cause whichever occurs first.
Overall Response Rate (ORR) | Measured up to 2 years after the last participant has enrolled in the study
  Overall response rate will be defined as the proportion of participants who achieve a partial remission or better.
Time to Tumor Progression (TTP) | Measured up to 2 years after the last participant has enrolled in the study
  Time to tumor progression is defined as the number of days from the date of study drug start to the date of the first documented disease progression or relapse.
Duration of Response (DOR) | Measured up to 2 years after the last participant has enrolled in the study
  Duration of response is defined as the number of days from the date of documented first response of partial remission or better to the date of documented disease progression/relapse or death due to the disease whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: John Hayslip, MD, Study Director — AbbVie
Locations (10):
- United States (10):
  - Site Reference ID/Investigator# 145677, Tucson, Arizona
  - Site Reference ID/Investigator# 147922, Chicago, Illinois
  - Site Reference ID/Investigator# 148562, Harvey, Illinois
  - Site Reference ID/Investigator# 148561, Goshen, Indiana
  - Site Reference ID/Investigator# 145674, Baltimore, Maryland
  - Site Reference ID/Investigator# 145145, Boston, Massachusetts
  - Site Reference ID/Investigator# 148010, Detroit, Michigan
  - Site Reference ID/Investigator# 147747, St Louis, Missouri
  - Site Reference ID/Investigator# 145146, Lebanon, New Hampshire
  - Site Reference ID/Investigator# 148559, Greenville, South Carolina